CLINICAL TRIAL: NCT04657926
Title: A Placebo-controlled, Double-blinded, Randomized, Trial Using a Combination of Apocynin and Paeonol (APPA) for the Treatment of Knee Osteoarthritis
Brief Title: A Trial of APPA in the Treatment of Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AKL Research and Development (Industry)
Collaborators: NBCD A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APPA-P2-1
Record Dates: First submitted 2020-11-30; First posted 2020-12-08 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — diadenosine pyrophosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APPA (Experimental): APPA, an oral combination of two isomers: 4-hydroxy-3-methoxyacetophenone (4H3MA) & 2-hydroxy-4-methoxyacetophenone (2H4MA) administered to 75 participants as 2 x 400mg capsules b.d. for 28 days
  .
  Interventions: Drug: APPA
- Placebo (Placebo Comparator): 2 capsules b.d. for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APPA — APPA, an oral combination of two isomers: 4-hydroxy-3-methoxyacetophenone (4H3MA) & 2-hydroxy-4-methoxyacetophenone (2H4MA).
  Arms: APPA
Drug: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
A placebo controlled study of APPA in 150 participants with Osteoarthritis of the knee

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel group, 4-week trial of a fixed-dose combination of apocynin and paeonol (APPA) administered orally twice daily versus placebo twice daily. Approximately 150 subjects will be randomized to one of the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to read and understand the language and content of the study material, understand the requirements for study visits, and is willing to provide information at the scheduled evaluations and appropriate written informed consent has been obtained.
2. Femorotibial osteoarthritis of the knee, according the American College of Rheumatology (ACR) clinical and radiographic criteria (Altman et al., 1986) (Appendix A).
3. Radiological OA grade 2 or 3 of the target knee, using the Kellgren-Lawrence method (Kellgren and Lawrence, 1957) as graded by central, independent reading of X-ray obtained during screening, or on a recent (within 6 months) X-ray image which fulfills the protocol specifications for reading.
4. Age between 40 years and 85 years at the time of screening, both included; of either sex.
5. Pain score rated on an 11-point numerical rating scale of the target knee of ≥ 20 and ≤ 45 out of 50 in response to the WOMAC pain sub-score (5 questions), at the time of screening and baseline. The subject should have undergone a washout-period of at least 5 half-lives of any analgesic medication before completing the screening and baseline questionnaires.
6. Women of child-bearing potential must use a highly effective method of contraception(please see Appendix B). Postmenopausal status is defined as being amenorrheic for at least 1 year prior to screening. Sexually active men with a female partner of childbearing potential must ensure that their female partner uses a highly effective method of contraception and agree to use condom from enrolment up to at least 3 months after the study end. Furthermore, male participants must agree not to donate sperm throughout the study and at least 3 months after he study end.
7. Knee pain in the target knee for 14 days of the preceding month (periarticular knee pain due to OA and not due to non-OA conditions such as bursitis, tendonitis, etc.) based on subject report.
8. Inadequate response to or intolerance to analgesics and/or non-steroidal anti-inflammatory drugs (NSAIDs) as reported by the subject

Exclusion Criteria:

1. Known or suspected hypersensitivity to or previous hypersensitivity reactions to APPA, or any of the excipients in the investigational product.
2. For women of childbearing potential:

   1. Pregnancy (i.e. positive pregnancy test at Screening) or breastfeeding
   2. Failure to agree to practice a highly effective method of contraception (see Appendix B), from enrolment up to at least 3 months after the study end.
3. For sexually active men with a female partner of childbearing potential: Failure to agree to ensure that their female partner uses a highly effective method of contraception, to agree to use condom (see Appendix B) from enrolment up to at least 3 months after the study end, and to agree not to donate sperm throughout the study and at least 3 months after the study end.
4. Intra-articular delivery of corticosteroids within 3 months or hyaluronic acid within 6 months of screening in the target knee or into any other joint within 30 days of screening.
5. Systemic corticosteroid treatment of more than 14 days during the past 6 months prior to screening.
6. Major surgery or arthroscopy of the target knee within the previous year prior to screening.
7. Planned surgery on either knee within the next 3 months.
8. Use of a currently unapproved investigational drug, device or biologic within 3 months prior to screening.
9. Presence of inflammatory arthritis, such as rheumatoid arthritis, psoriatic arthritis, polymyalgia rheumatica, gout or pseudogout with history of clinical attacks.
10. Current malignancy or treatment for malignancy within the past five years, with the exception of treated non-melanoma skin cancer, unless affecting the target knee area, or carcinoma in situ events.
11. Any other abnormal laboratory results or significant medical conditions that the Investigator believes should preclude the subject's participation in the trial.
12. Prior septic arthritis of the target knee.
13. Known osteoarthritis of the hip(s) if pain in either or both hip(s) exceeds that of the target knee using the WOMAC Hip Pain sub-score for that hip at the time of screening
14. Presence of significant radicular back pain, as reported by the subject.
15. Presence of severe pain in either knee, defined as > 45 out of 50 in response to the WOMAC pain sub-score (5 questions), at the time of screening or baseline, regardless of the eligibility of the contralateral knee.
16. Body Mass Index > 40.0 kg/m2.
17. Estimated glomerular filtration rate < 30 mL/min using the Modification of Diet in Renal Disease (MDRD) method.
18. Substantial use of moderate or higher strength opioid medication for the treatment of pain within 6 weeks before the screening visit, as evaluated by the investigator.
19. Use of duloxetine, pregabalin, or gabapentin within 4 weeks before the baseline visit.
20. History of alcohol or drug abuse within the past 5 years prior to randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
WOMAC pain score | 28 days
  change from baseline in WOMAC pain sub-score of the target knee as evaluated at week 4.

SECONDARY OUTCOMES:
Changes from baseline in WOMAC total score and the WOMAC function and stiffness scores at week 4 | 28 days
Changes from baseline in constant, intermittent and total OA pain assessed by ICOAP scores at week 4 Changes from baseline in constant, intermittent and total OA pain assessed by ICOAP scores at week 4 | 28 days
Changes from baseline in WOMAC pain weight-bearing score (questions 1, 2, and 5) and non-weight bearing score (questions 3 and 4) at week 4 | 28 days
Changes from baseline in physical function assessed by the 20 Meter Walk Test gait speed at week 4 | 28 days
Change from baseline in the weekly mean of the average daily pain intensity at Week 4 | 28 days
Area-under-effect curves of the weekly mean of the average daily pain intensity at Week 4 | 28 days
OMERACT-OARSI responder rate at week 4 | 28 days
Total dose of rescue medication calculated as the sum of tablets used, based on pill counts | 28 days
Time between baseline and first use of rescue medication | 28 days
Changes from baseline in the Patient Global Assessment (PGA) score at week 4 | 28 days
Changes from baseline in quality of life assessed by the EQ5D at week 4 | 28 days
Safety | 28 days
  Nature, incidence and severity of AEs. Changes in laboratory safety parameters, vital signs, 12-lead ECG parameters, and weight

OTHER OUTCOMES:
Changes in serum and urine biomarkers of joint tissue turnover | 28 days
  At baseline, and during the trial, serum and urine will be collected, for measurement of biomarkers reflecting collagen- and proteoglycan turnover
Time to achieve a clinically relevant pain reduction defined as a decrease from baseline of at least 1 points out of 10 in the 11-point average of daily pain score | 28 days
Time to achieve "moderate improvement" and time to achieve "high improvement" in OMERACT-OARSI response | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Asger Bihlet, Study Director — Nordic Bioscience Clinical Development
Locations (1):
- Sanos Clinic, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yao Q, Wei T, Qiu H, Cai Y, Yuan L, Liu X, Li X. Epigenetic Effects of Natural Products in Inflammatory Diseases: Recent Findings. Phytother Res. 2025 Jan;39(1):90-137. doi: 10.1002/ptr.8364. Epub 2024 Nov 8. PMID 39513382